CLINICAL TRIAL: NCT04881331
Title: Intraoperative Tissue Identification by Analyzing Surgical Smoke
Acronym: SurgiNose
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Niku Oksala, Professor of Surgery, Chief physician, Tampere University Hospital
Other Study IDs: R17096
Record Dates: First submitted 2021-05-07; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Analysis of electrosurgical smoke. — Patients undergo standard of care surgical removal of the malignant breast tumor. Electrosurgical knife is used to cut tissues according to standard practice. Fraction of the surgical smoke is captured for analysis and video record of the point of view of the surgeon is captured with a head-mounted camera.

SUMMARY:
SurgiNose is a single-center, non-randomized feasibility study aiming to evaluate the feasibility of intraoperative tissue analysis using differential mobility of surgical smoke generated with electrocautery.

Patients receive standard-of-care breast conserving surgery.

DETAILED DESCRIPTION:
The increasing number of breast cancer survivors and their longevity has emphasized the importance of aesthetic and functional outcomes of cancer surgery and increased pressure for the surgical treatment to achieve negative margins with minimal removal of healthy tissue.

Surgical smoke has been successfully utilized in tissue identification in laboratory conditions by using a system based on differential mobility spectrometry (DMS) that could provide a seamless margin assessment method.

In this study, a DMS-based tissue smoke analysis system will be used intraoperatively in 20 breast cancer surgeries to assess its feasibility in tissue identification. The effect of the system on complications and duration of surgeries is also studied. The surgeries are recorded with a head-worn camera system for visual annotation of the operated tissue types to enable classification of the measurement files by supervised learning.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary malignancy of the breast

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological female
Study Population: Patients undergoing breast conserving surgery for histologically confirmed malignancy of the breast. There is no upper limit for participation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Discrimination rate of healthy tissue types encountered during surgery | During the procedure
  The device records a molecular spectrum of the surgical smoke every time the device is activated. The tissues are annotated using head-mounted camera that records video footage from the viewpoint of the surgeon.
  The primary outcome of the the study is the ability of the device to correctly classify healthy tissues that are encountered during breast surgery including fat tissue, glandular tissue, connective tissue, muscle tissue, dermis. The accuracy is cross-validated using leave-one-out cross-validation and is reported as correct classification rate (CCR) %.

SECONDARY OUTCOMES:
Surgical time | During the procedure
  The duration of surgical procedures when the device is used. Institutional average procedure duration is used for comparison.
Complications | 30 days after surgery.
  Complications of surgery in the follow-up period of 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- TAYS Hatanpää, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutinen M, Kontunen A, Karjalainen M, Kiiski J, Hannus J, Tolonen T, Roine A, Oksala N. Identification of breast tumors from diathermy smoke by differential ion mobility spectrometry. Eur J Surg Oncol. 2019 Feb;45(2):141-146. doi: 10.1016/j.ejso.2018.09.005. Epub 2018 Oct 15. PMID 30366874